CLINICAL TRIAL: NCT04247308
Title: Multi-modal Stimulations on Neuromotor Responses Among the Hospitalised Preterm Infants
Brief Title: Multi Modal Stimulations in Pre-term Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/IEC/1566; U1111-1236-9478 (Other: UTN by WHO International Clinical Trials Registry Platform)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Preterm Birth; Infant, Premature, Diseases
Keywords: Preterm; Neonate; Multi-modal stimulation
MeSH Terms: conditions — Premature Birth; Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: Two group pre-test post-test design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Sensory stimulations (ATVV) will be consisting of Soft lullaby between of 30-40 dB for Auditory, Gentle stroking massage in supine position(upper and lower limb)for Tactile, Visual Stimulations with Black and white card (distance of 8-10 in), gentle rocking (vertical and horizontal direction) for the stimulation of vestibular system and oral stimulation including stocking cheeks, lips, jaw and tongue, rubbing gum.Each stimulation will be given for 3 minutes.
  Movement therapy will include: Guided range of motion: flexion-extension movements of lower limb (bicycle riding pattern). Hand should be placed around knee joint. Care must be taken as PI consist the cartilaginous joints at wrist and ankle. Anti gravity movements in prone (neck and spinal extension), Anti gravity movements in sitting (supported) and Upright positioning for 3min each
  Interventions: Other: Sensory Stimulation; Other: Movement therapy
- control group (Active Comparator): receives routine care from the nursing team as well as daily maternal care, such as being held in the mother's arms
  Interventions: Other: Routine hospital care

INTERVENTIONS:
Other: Sensory Stimulation — Auditory, tactile, visual, vestibular and oro motor stimulation
  Arms: experimental group
Other: Movement therapy — Passive range of movements, antigravity movements in prone and supine
  Arms: experimental group
Other: Routine hospital care — Maintaining the vitals
  Arms: control group

SUMMARY:
A total of 56 neonates with LBW will recruited by the convenience sampling to participate in this two group pre-test post-test, single blinded randomized clinical study. After the demographics, recruited NLBW will be randomly divided into two groups, group A and group B with block randomization. There will be four blocks, with the matrix design of 4X14 here 14 being rows. Each block contained 4 chits (2 chits for each group), totalling 56. The subjects will be allotted to the group based on the randomly chosen chit by their parents. Once the block will be allotted, next row block was opened. Thus, equal number of NLBW will be assigned to each group over time.

Group A will be receiving multimodal sensory and kinesthetic stimulation (MSKS) and Group B will be receiving regular lifesaving hospital care. Group A will receive the interventions for 2 weeks period, totalling 10 sessions. Each session will last for 30 minutes duration.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born between 28 and 36 week of gestation
2. Birth weight ranging from 1000-2500 g.
3. Medically stable preterm infants

Exclusion Criteria:

1. Medically unstable preterm infants.
2. Infants with congenital anomalies, congenital infections and central nervous system injury

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Infant Neurological International Battery | Change from baseline and 2 weeks
  Infant Neurological International Battery (INFANIB), the minimum and maximum values are 14 and 70 respectively, and higher scores mean a better outcome. Scores less than and equal to 48 is abnormal while greater than and equal to 66 means normal.

CONTACTS AND LOCATIONS:
Overall Officials: Vencita P Aranha, MPT, (PhD), Principal Investigator — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, MM(DU)
Locations (1):
- Neonatal Intensive Care Unit, Maharishi Markandeshwar Hospital, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Publication in Peer-Reviewed Indexed Journals
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the end of the study
Access Criteria: Mendeley data
URL: http://data.mendeley.com/datasets/k4j689jfwj/2

REFERENCES:
- [Background] Aranha VP, Chahal A, Bhardwaj AK. Neonatal aquatic physiotherapy in neonatal intensive care units: A scoping review. J Neonatal Perinatal Med. 2022;15(2):229-235. doi: 10.3233/NPM-210858. PMID 34719445
- [Result] Aranha VP, Chahal A, Bhardwaj AK. Short-term effects of multimodal stimulation on neuromotor behaviour and neonatal pain among hospitalized preterm infants: A feasibility, non-blinded randomized controlled trial. J Neonatal Perinatal Med. 2023;16(2):325-337. doi: 10.3233/NPM-210889. PMID 34864695
- Available data/document: Individual Participant Data Set: Mendeley Data — http://data.mendeley.com/datasets/k4j689jfwj/2 — Contains 56 Preterm Infants data which includes, gestational age, chronological age, corrected gestational age, sex, birth weight, birth length, birth occipitofrontal circumference (OFC), APGAR at 1-min, and APGAR at 5-min, pre-post intervention (5 days) changes of weight, length, OFC, INFANIB (Infant Neurological International Battery) and NIPS (Neonatal Infant Pain Scale).